CLINICAL TRIAL: NCT00081211
Title: A Phase I Study Of PV701 In Patients With Head And Neck Squamous Cell Carcinoma
Brief Title: Intratumoral PV701 in Treating Patients With Advanced or Recurrent Unresectable Squamous Cell Carcinoma of the Head and Neck
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Administratively complete.
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02723; 12157B; N01CM17102 (NIH); CDR0000360664 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2004-04-07; First posted 2004-04-08 (Estimated); Last update posted 2013-01-24 (Estimated); Status verified 2013-01

CONDITIONS: Recurrent Salivary Gland Cancer; Recurrent Squamous Cell Carcinoma of the Hypopharynx; Recurrent Squamous Cell Carcinoma of the Larynx; Recurrent Squamous Cell Carcinoma of the Lip and Oral Cavity; Recurrent Squamous Cell Carcinoma of the Nasopharynx; Recurrent Squamous Cell Carcinoma of the Oropharynx; Recurrent Squamous Cell Carcinoma of the Paranasal Sinus and Nasal Cavity; Salivary Gland Squamous Cell Carcinoma; Stage III Salivary Gland Cancer; Stage III Squamous Cell Carcinoma of the Hypopharynx; Stage III Squamous Cell Carcinoma of the Larynx; Stage III Squamous Cell Carcinoma of the Lip and Oral Cavity; Stage III Squamous Cell Carcinoma of the Nasopharynx; Stage III Squamous Cell Carcinoma of the Oropharynx; Stage III Squamous Cell Carcinoma of the Paranasal Sinus and Nasal Cavity; Stage IV Salivary Gland Cancer; Stage IV Squamous Cell Carcinoma of the Hypopharynx; Stage IV Squamous Cell Carcinoma of the Larynx; Stage IV Squamous Cell Carcinoma of the Lip and Oral Cavity; Stage IV Squamous Cell Carcinoma of the Nasopharynx; Stage IV Squamous Cell Carcinoma of the Oropharynx; Stage IV Squamous Cell Carcinoma of the Paranasal Sinus and Nasal Cavity
MeSH Terms: conditions — Salivary Gland Neoplasms; Squamous Cell Carcinoma of Head and Neck

ARMS (1):
- Treatment (PV701) (Experimental): Patients receive intratumoral PV701 once weekly for 3 weeks. Courses repeat every 6 weeks in the absence of disease progression or unacceptable toxicity. Cohorts of 3-6 patients receive escalating doses of PV701 until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity. Once the MTD is determined, at least 6 evaluable patients are treated at that dose.
  Interventions: Biological: PV701

INTERVENTIONS:
Biological: PV701 — Given intratumorally

SUMMARY:
Phase I trial to study the effectiveness of intratumoral (in the tumor) PV701 in treating patients who have advanced or recurrent unresectable squamous cell carcinoma (cancer) of the head and neck. Vaccines made from a specially-modified virus such as PV701 may make the body build an immune response to kill tumor cells while leaving normal cells undamaged. Injecting PV701 directly into the tumor may cause a stronger immune response and kill more tumor cells

DETAILED DESCRIPTION:
OBJECTIVES:

I. Determine the maximum tolerated dose (MTD) of PV701 administered by direct intratumoral injection in patients with advanced or recurrent unresectable squamous cell carcinoma of the head and neck.

II. Determine the toxicity of intratumoral PV701 in these patients. III. Determine response rate and time to progression at the injection site in patients treated with this drug.

OUTLINE: This is a dose-escalation study. Patients receive intratumoral PV701 once weekly for 3 weeks. Courses repeat every 6 weeks in the absence of disease progression or unacceptable toxicity. Cohorts of 3-6 patients receive escalating doses of PV701 until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity. Once the MTD is determined, at least 6 evaluable patients are treated at that dose.

PROJECTED ACCRUAL: A maximum of 30 patients will be accrued for this study within 6-10 months.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed squamous cell carcinoma of the head and neck

  * Locally advanced or recurrent disease
  * Distant metastases in addition to locally advanced disease acceptable
* Not amenable to available standard treatment or palliative measures
* At least one target lesion accessible for intratumoral injection, less than 4 cm, and not situated near an airway or major artery
* Tumor volume(s) must be large enough to receive injection
* No known brain metastases
* Performance status - ECOG 0-2
* More than 3 months
* WBC >= 3,000/mm^3
* Hemoglobin > 10 g/dL (transfusion permitted)
* Platelet count >= 100,000/mm^3
* Bilirubin < 2 times upper limit of normal (ULN)
* AST/ALT =< 2.5 times ULN
* Creatinine < 2.5 mg/dL
* No uncontrolled symptomatic congestive heart failure
* No unstable angina pectoris
* No cardiac arrhythmia
* No history of significantly compromised pulmonary function (i.e. FEV_1 < 50% of predicted) or decreased oxygen saturation of < 95% on room air
* No history of allergy to eggs or egg-based or chicken embryo-based vaccines
* No frequent contact with immunocompromised individuals
* No ongoing or active infection
* No psychiatric illness or social situation that would preclude study compliance
* No history of diabetes mellitus requiring oral hypoglycemic agents or insulin
* No HIV-positive patients receiving combination antiretroviral therapy
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* More than 4 weeks since prior chemotherapy and recovered
* More than 4 weeks since prior radiotherapy and recovered
* More than 4 weeks since prior surgery and recovered
* No other concurrent investigational agents or commercial agents or therapies for treatment of malignancy
* No concurrent antiviral therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2004-04; Primary Completion 2004-07 (Actual)

PRIMARY OUTCOMES:
Maximum-tolerated dose (MTD) of PV701 based on the incidence of dose-limiting toxicity (DLT) as assessed by NCI Common Terminology Criteria for Adverse Events (CTCAE) version 3.0 | 3 weeks

SECONDARY OUTCOMES:
Toxicity as assessed by NCI CTCAE version 3.0 | Up to 12 weeks
Response (complete and partial) rate according to Response Evaluation Criteria in Solid Tumors (RECIST) Committee | Up to 12 weeks
  Descriptive statistics will be generated for each group.
Time to progression according to RECIST | From the time of study entry until tumor growth is determined by physical exam or by radiographic imaging, assessed up to 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: David Gustin, Principal Investigator — University of Chicago Comprehensive Cancer Center
Locations (1):
- University of Chicago Comprehensive Cancer Center, Chicago, Illinois, United States